CLINICAL TRIAL: NCT03496324
Title: A Randomised, Single-dose, 4-way Crossover, Open-label, Pharmacokinetic Study Comparing a 4% (w/v) Suspension of Ibuprofen With a Reference 2% (w/v) Suspension of Ibuprofen in the Fed and Fasted States.
Brief Title: Ibuprofen 4% (w/v) Pivotal Bioequivalence Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: RB7-UK-1509; 2015-003894-13 (EudraCT Number)
Record Dates: First submitted 2018-04-05; First posted 2018-04-12 (Actual); Results first posted 2019-06-05 (Actual); Last update posted 2019-06-05 (Actual); Status verified 2019-02

CONDITIONS: Bioequivalence of the Test Formulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Test (fed): Nurofen for Children (Active Comparator): Nurofen for Children® 400 mg/10 ml by mouth under fed condition
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Interventions: Drug: Nurofen for Children®
- Test (fasted): Nurofen for Children (Active Comparator): Nurofen for Children® 400 mg/10 ml by mouth under fasted condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Interventions: Drug: Nurofen for Children®
- Reference (fed): Algifor Junior (Experimental): Algifor® Junior 400 mg/20 ml by mouth under fed condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Interventions: Drug: Algifor® Junior
- Reference (fasted): Algifor Junior (Experimental): Algifor® Junior 400 mg/20 ml by mouth under fasted condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Interventions: Drug: Algifor® Junior

INTERVENTIONS:
Drug: Nurofen for Children® — Nurofen for Children® 400 mg/10 ml
  Other Names: NfC®
  Arms: Test (fasted): Nurofen for Children; Test (fed): Nurofen for Children
Drug: Algifor® Junior — Algifor® Junior 400 mg/20 ml
  Other Names: Ibuprofen oral suspension
  Arms: Reference (fasted): Algifor Junior; Reference (fed): Algifor Junior

SUMMARY:
Bioequivalence evaluation of Nurofen for Children® with reference formulation of Algifor® Junior by determining and comparing the rate and extent of absorption in both fed and fasted states

ELIGIBILITY:
Inclusion Criteria:

1. Subjects who had given written informed consent.
2. Age: ≥18 years ≤50 years.
3. Sex: Male or female subjects who were eligible for entry.
4. Female subject of childbearing potential with a negative pregnancy test at the screening visit and who were willing to use an effective method of contraception, if applicable (unless of non-childbearing potential or where abstaining from sexual intercourse was in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after the final dose of Investigational Medicinal Product (IMP). Effective forms of contraception included: established use of oral, injected or implanted hormonal methods of contraception, placement of an intrauterine device (IUD) or intrauterine system (IUS), barrier methods of contraception: condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, male sterilisation (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate).
5. Female subject of non-child bearing potential with negative pregnancy test at the screening visit. For the purposes of this study, this was defined as the subject being amenorrheic for at least 12 consecutive months or at least 4 months post-surgical sterilisation (including bilateral fallopian tube ligation or bilateral oophorectomy with or without hysterectomy). Menopausal status was confirmed by demonstrating at screening that levels of follicle stimulating hormone (FSH) fell within the respective pathology reference range. In the event a subject's menopause status had been clearly established (for example, the subject indicated she had been amenorrheic for 10 years), but FSH levels were not consistent with a post-menopausal condition, determination of subject eligibility was at the discretion of the Principal Investigator following consultation with the Sponsor's Responsible Physician.
6. Male subject willing to use an effective method of contraception, if applicable (unless anatomically sterile or where abstaining from sexual intercourse in line with the preferred and usual lifestyle of the subject) from first dose until 3 months after the final dose of IMP.
7. Healthy subjects as determined by past medical history, physical examination, vital signs, electrocardiogram (ECG), and laboratory tests at screening.
8. Healthy subjects with a body mass index (BMI) of ≥20 and ≤27 kg/m2.

Exclusion Criteria:

1. Pregnant or lactating females.
2. A history and/or presence of significant disease of any body system, including psychiatric disorders as specified in Chapter 5 of the International Classification of Diseases (ICD) 10.
3. Any condition that may have interfered with the absorption, distribution, metabolism or excretion of drugs.
4. A history of allergy or intolerance (including angioedema, urticaria, bronchospasm and rhinitis) related to treatment with ibuprofen, aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), or the excipients of the formulations.
5. A history of or active peptic or duodenal ulcers or gastrointestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
6. A history of frequent dyspepsia, e.g. heartburn or indigestion.
7. A history of migraine.
8. Users of nicotine products i.e. current smokers and ex-smokers who had smoked within the 6 months prior to dosing with the study medication or users of cigarette replacements (e.g. e-cigarettes, nicotine patches or gums).
9. A history of substance abuse (including alcohol).
10. High consumption of stimulating drinks (coffee, tea, cola, energy drinks etc. total caffeine intake per day above 300 mg (1 cup of coffee equated to 50 mg)).
11. Those with positive screen/test for drugs of abuse including alcohol on any occasion throughout the study.
12. Ingestion of a prescribed drug at any time in the 14 days before dosing with study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers during the previous month (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc.).
13. Ingestion of an over-the-counter preparation within 7 days before dosing with study medication, including herbal medications, vitamin/fish oil supplements, ibuprofen and other NSAID.
14. Donation of blood in quantity >400 mL, e.g., to the blood transfusion service in the previous 12 weeks before enrolment into the study.
15. Known human immune deficiency virus (HIV) positive status, or a positive viral serology screen.
16. Topical use of ibuprofen within 7 days before dosing with IMP.
17. Those previously randomized into this study.
18. Employee at study site.
19. Partner or first degree relative of the Investigator.
20. Those who have participated in a clinical trial in the previous 12 weeks.
21. Those unable, in the opinion of the Investigator, to comply fully with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2016-05-06 (Actual); Study Completion 2016-05-06 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted in single-site in the United Kingdom.
Pre-assignment Details: Total 71 subjects were screened. Of these, 38 subjects were screen failures, 2 were withdrew consent, 7 were reserve subjects. Subjects randomized were 24.
Groups:
- Sequence 1-BACD: Test (Fed) - Nurofen for Children: B = Nurofen for Children® 400 mg/10 ml (Test fasted)
  A = Nurofen for Children® 400 mg/10 ml (Test fed)
  C = Algifor® Junior 400 mg/20 ml (Reference fed)
  D = Algifor® Junior 400 mg/20 ml (Reference fasted)
- Sequence 2-DCAB: Test (Fasted) - Nurofen for Children: D = Algifor® Junior 400 mg/20 ml (Reference fasted)
  C = Algifor® Junior 400 mg/20 ml (Reference fed)
  A = Nurofen for Children® 400 mg/10 ml (Test fed)
  B = Nurofen for Children® 400 mg/10 ml (Test fasted)
- Sequence 3-ADBC: Reference (Fed) - Algifor Junior: A = Nurofen for Children® 400 mg/10 ml (Test fed)
  D = Algifor® Junior 400 mg/20 ml (Reference fasted)
  B = Nurofen for Children® 400 mg/10 ml (Test fasted)
  C = Algifor® Junior 400 mg/20 ml (Reference fed)
- Sequence 4-CBDA: Reference (Fasted) - Algifor Junior: C = Algifor® Junior 400 mg/20 ml (Reference fed)
  B = Nurofen for Children® 400 mg/10 ml (Test fasted)
  D = Algifor® Junior 400 mg/20 ml (Reference fasted)
  A = Nurofen for Children® 400 mg/10 ml (Test fed)
Period: Period 1
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 1: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 2: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 3: Washout (3 to 7 Days)
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0
Period: Period 7: Period 4
Arm/Group | Sequence 1-BACD: Test (Fed) - Nurofen for Children | Sequence 2-DCAB: Test (Fasted) - Nurofen for Children | Sequence 3-ADBC: Reference (Fed) - Algifor Junior | Sequence 4-CBDA: Reference (Fasted) - Algifor Junior
Started | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Nurofen for Children® 400 mg/10 mL single-oral dose under fasted and fed conditions.
  Algifor® Junior 400 mg/20 mL single-oral dose under fasted and fed conditions.
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (8.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 22
  More than one race | 0
  Unknown or Not Reported | 2
Weight [Mean (Standard Deviation); unit: kg] | 68.68 (11.506)
Height [Mean (Standard Deviation); unit: meter] | 1.692 (0.0935)
Body Mass Index [Mean (Standard Deviation); unit: kg/m²] | 23.82 (2.037)

OUTCOME MEASURES:

1. Primary Outcome: Maximum Plasma Concentration (Cmax) of Ibuprofen
Description: One Subject in Period 3 Reference (fasted) was not included in PK Parameter Summary Set as per statistical analysis plan (SAP) Population definitions.
Time Frame: Pre-dose (Day -1), 10, 15, 20, 30, 40, 50, 60, 70, 80, 90, 105, 120, 180, 240, 360, 480 and 720 minutes (Day 0) post-dose
Population: Pharmacokinetics (PK) Parameter Summary Set population: All subjects from the PK dataset with evaluable PK parameters for each treatment period. (PK Dataset: All subjects from the safety population with evaluable plasma concentrations).
Measure: Mean (Standard Deviation); unit: μg/ml
Groups:
- Test (Fasted): Nurofen for Children: Nurofen for Children® 400 mg/10 ml by mouth under fasted condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Nurofen for Children®: Nurofen for Children® 400 mg/10 ml
- Test (Fed): Nurofen for Children: Nurofen for Children® 400 mg/10 ml by mouth under fed condition
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Nurofen for Children®: Nurofen for Children® 400 mg/10 ml
- Reference (Fasted): Algifor Junior: Algifor® Junior 400 mg/20 ml by mouth under fasted condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Algifor® Junior: Algifor® Junior 400 mg/20 ml
- Reference (Fed): Algifor Junior: Algifor® Junior 400 mg/20 ml by mouth under fed condition.
  Subjects participated in Treatment Sequence: BACD, DCAB, ADBC and CBDA.
  Algifor® Junior: Algifor® Junior 400 mg/20 ml
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
μg/ml | 38.503 (7.5696) | 25.162 (6.9668) | 33.843 (3.7858) | 26.432 (6.129)
Statistical Analysis 1: Comparison: Test (Fed): Nurofen for Children vs Reference (Fed): Algifor Junior; Test type: Equivalence — Bioequivalence was demonstrated between NfC® and Algifor® Junior if each 90% confidence interval (CI) (rounded to 2 decimal places) for the ratio between least square geometric means (test / reference) lay within 80% and 125% for Cmax; Geometric Least Square Mean = 94.19, 90% CI 2-sided [85.81 to 103.38], Standard Error of Mean 18.9
Statistical Analysis 2: Comparison: Test (Fasted): Nurofen for Children vs Reference (Fasted): Algifor Junior; Test type: Equivalence — Bioequivalence was demonstrated between NfC® and Algifor® Junior if each 90% CI (rounded to 2 decimal places) for the ratio between least square geometric means (test / reference) lay within 80% and 125% for Cmax; Geometric Least Square Mean = 111.66, 90% CI 2-sided [103.84 to 120.07], Standard Error of Mean 14.3

2. Primary Outcome: Area Under Plasma Concentration-time Curve From Administration to the Last Quantifiable Concentration at Time t (AUC0-t) of Ibuprofen
Time Frame: as for outcome 1
Population: PK Parameter Summary set population. One Subject in Period 3 Reference (fasted) was not included in PK Parameter Summary Set as per statistical analysis plan (SAP) Population definitions.
Measure: Mean (Standard Deviation); unit: min*μg/mL
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
min*μg/mL | 6169.662 (1199.1785) | 5754.831 (1056.5014) | 5960.054 (832.1342) | 5482.340 (827.2913)
Statistical Analysis 1: Comparison: Test (Fasted): Nurofen for Children vs Reference (Fasted): Algifor Junior; Test type: Equivalence — Bioequivalence was demonstrated between NfC® and Algifor® Junior if each 90% CI (rounded to 2 decimal places) for the ratio between least square geometric means (test / reference) lay within 80% and 125% for AUC0-t; Geometric Least Square Mean = 101.57, 90% CI 2-sided [96.28 to 107.16], Standard Error of Mean 10.5
Statistical Analysis 2: Comparison: Test (Fed): Nurofen for Children vs Reference (Fed): Algifor Junior; Test type: Equivalence — [test comment as in outcome 2, analysis 1]; Geometric Least Square Mean = 104.47, 90% CI 2-sided [101.4 to 107.63], Standard Error of Mean 6

3. Secondary Outcome: Elimination Rate Constant (Kel) of Ibuprofen
Description: Kel was calculated as the absolute value of the log-linear regression slope of the elimination phase (logged) over time (linear) using the post Cmax concentrations [at least 3 non-below the limit of quantification (BLQ)] that maximized the adjusted R2.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/min
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
1/min | 0.00646 (0.000763) | 0.00532 (0.00119) | 0.00668 (0.000763) | 0.00577 (0.000865)

4. Secondary Outcome: Area Under Plasma Concentration-time Curve From Administration to Infinity (AUC0-inf) of Ibuprofen
Description: AUC0-inf was calculated as AUC0-t + (Ct/Kel) where Ct was the last quantifiable concentration at time t.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min*μg/mL
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
min*μg/mL | 6255.821 (1229.6414) | 5982.084 (1118.9361) | 6032.841 (843.8379) | 5609.733 (862.2304)

5. Secondary Outcome: Ratio of AUC0-t/AUC0-inf (AUCR)
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
Ratio | 0.987 (0.0066) | 0.963 (0.0384) | 0.988 (0.0052) | 0.978 (0.0142)

6. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Ibuprofen
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
min | 60.4 (43.59) | 65.8 (24.79) | 65 (33.81) | 74.9 (42.66)

7. Secondary Outcome: Plasma Concentration Half-life (T1/2) of Ibuprofen
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: min
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 23 | 24
min | 108.854 (13.1303) | 138.894 (41.0392) | 104.975 (11.6362) | 122.752 (19.338)

8. Secondary Outcome: Number of Subjects With Treatment Emergent Adverse Events (TEAEs)
Description: Mild = Adverse event (AE) did not limit usual activities; subject may have experienced slight discomfort.
  Moderate = AE resulted in some limitation of usual activities; subject may have experienced significant discomfort.
  Severe = AE resulted in an inability to carry out usual activities; subject may have experienced intolerable discomfort/pain.
  Unassessable/Unclassified = Insufficient information to be able to make an assessment Conditional/ Unclassified = Insufficient information to make an assessment at present Unrelated = No possibility that the AE was caused by the IMP Unlikely = Slight, but remote, chance that the AE was caused by the IMP, but the balance of judgment was that it was most likely not due to the investigational medicinal product (IMP).
  Possible = Reasonable suspicion that the AE was caused by the IMP Probable = Most likely that the AE was caused by the IMP Certain = AE was definitely caused by the IMP
Time Frame: Up to Day 7 (follow-up)
Population: Safety population: All subjects who received at least 1 dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
Number analyzed (Participants) | 24 | 24 | 24 | 24
Participants
  Treatment Emergent Adverse Event (TEAE) | 3 | 1 | 1 | 0
  Serious TEAE | 0 | 0 | 0 | 0
  TEAE Leading to Withdrawal | 0 | 0 | 0 | 0
  TEAE by severity: Mild | 3 | 1 | 1 | 0
  TEAE by severity: Moderate | 0 | 0 | 0 | 0
  TEAE by severity: Severe | 0 | 0 | 0 | 0
  Relationship to IMP - Certain | 0 | 0 | 0 | 0
  Relationship to IMP - Probable | 0 | 0 | 0 | 0
  Relationship to IMP - Possible | 0 | 0 | 0 | 0
  Relationship to IMP - Unlikely | 0 | 0 | 0 | 0
  Relationship to IMP - Unrelated | 3 | 1 | 1 | 0
  Relationship to IMP - Conditional/Unclassified | 0 | 0 | 0 | 0
  Relationship to IMP - Unassessable/Unclassifiable | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Day 7 (Follow-up)
Arm/Group | Test (Fasted): Nurofen for Children | Test (Fed): Nurofen for Children | Reference (Fasted): Algifor Junior | Reference (Fed): Algifor Junior
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 1/24 | 1/24 | 0/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Fasted): Nurofen for Children (N=24) | Test (Fed): Nurofen for Children (N=24) | Reference (Fasted): Algifor Junior (N=24) | Reference (Fed): Algifor Junior (N=24)
Headache (Nervous system disorders) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No